CLINICAL TRIAL: NCT06386562
Title: Step by Step - Pilot Study of an Internet-based Parenting Program for Aggressive, Disruptive Behavior in Children and Adolescents
Brief Title: Pilot Study of an Internet-based Parenting Program for Child Disruptive Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Pia Enebrink, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-07489-01
Record Dates: First submitted 2024-04-08; First posted 2024-04-26 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Child Behavior Problem; Disruptive Behavior; Oppositional Defiant Disorder; Conduct Problems; Parent-Child Relations
Keywords: Disruptive Behavior; Child Behavior Problem; Parenting; Internet-based parent training
MeSH Terms: conditions — Problem Behavior; Oppositional Defiant Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based parenting program (Active Comparator): Internet-based parenting program with weekly parental support from a family guide (psychologist) via a chat function integrated into the program. The program consists of a brief introducing module and 5 modules conducted over 5-7 weeks. Parents work independently with material online and receive support from the family guide through chat/text messages in the program.
  Interventions: Behavioral: Family Check-up and Cognitive behavior therapy online: a Swedish internet-based parenting program
- Internet-based parenting program with additional parental support through digital/phone meetings (Experimental): The same internet-based parenting program with weekly parental support from a family guide (psychologist) via a chat function integrated into the program. The addition is three 10-15 minutes long digital/phone meetings between the family guide and the parent.
  Interventions: Behavioral: Family Check-up and Cognitive behavior therapy online: a Swedish internet-based parenting program with additional parental support

INTERVENTIONS:
Behavioral: Family Check-up and Cognitive behavior therapy online: a Swedish internet-based parenting program — The internet-based parenting support program is based on social learning theory. A foundation is the Family Check-up program (FCU), which includes approaches from motivational interviewing (MI). The parenting support is also based on similar CBT-parenting strategies as in other evaluated face-to-face CBT-parenting support programs (e.g., Comet) as well as internet-based programs (e.g., iComet; ParentWeb).
  Arms: Internet-based parenting program
Behavioral: Family Check-up and Cognitive behavior therapy online: a Swedish internet-based parenting program with additional parental support — The internet-based parenting program includes the same contents and chat-function as in the other condition. The focus for the digital/phone meetings is to explore potential questions, problem-solve around potential challenges, and motivate parents to practice strategies and complete modules.
  Arms: Internet-based parenting program with additional parental support through digital/phone meetings

SUMMARY:
The goal of this pilot randomized controlled trial is to learn about effects and experiences of an internet-based parenting program for parents of children and adolescents with behavioral problems (e.g., aggressive or defiant behavior).

The main questions the study aims to answer are:

* What are the preliminary effects of the internet-based parenting program?
* What is the level of parents' engagement in the parenting program?
* How do parents perceive the program?

Families will be randomized to a version of an internet-based parenting program with support provided from family guides (psychologists) through chat messages in the program, or to the same internet-based parenting program with additional phone/digital support-meetings. Parents will answer quantitative measurements questions before, during, and after treatment. Parents will also be asked to participate in a qualitative interview after the program. Both within and between group comparisons will be conducted to see if there are trends within each arm and differences between the two types of support.

DETAILED DESCRIPTION:
BACKGROUND:

Some children with behavior problems (e.g., aggressive and defiant behaviors) are at elevated risk for continued behavioral problems, and for developing more serious forms of antisocial behaviors as well as difficulties with peers, school and mental health issues. Early and effective interventions are needed to reduce the risk of behavioral problems escalating over time.

Parenting programs can be a first intervention for parents with children under 12 years old with oppositional defiant disorder or conduct disorder, or for parents of teenagers with less severe behavioral problems. Several parenting programs that show effectiveness in addressing behavioral problems are based on social learning theory and Cognitive Behavioral Therapy (CBT). One aim of parenting programs is to reduce negative interactions between parents and children (e.g., inconsistent, strict, and insensitive parenting) and to increase positive interactions (e.g., engagement, showing support, and encouragement). Examples of evaluated parenting programs for behavioral problems include Family Check-Up (FCU), The Incredible Years, and the Swedish parenting program Comet.

Generally, internet-based interventions have become increasingly available as a treatment option for families. These have the advantage of being easily accessible, possible to go through at a convenient time, reaching people in areas where certain interventions are not available, and can be provided at a low cost. The internet-based models often include some form of support from a therapist/family guide who assists the parents. There are several promising internet-based parenting programs for parents of children with behavioral problems. In Sweden, the internet-based parenting support iComet for parents of children aged 3-12 years with behavior problems has been developed, based on the Swedish face-to-face parenting program Comet, as well as the ParentWeb for parents of teenagers, targeting parents of youth with subclinical levels of behavior problems. However, there are few internet-based parenting programs for parents of school-age children and adolescents with early signs of behavior problems.

PURPOSE AND RESEARCH QUESTIONS:

The purpose of the present project is to conduct a first evaluation of a newly developed, internet-based parenting program based on the FCU and CBT strategies, targeting parents of children between 8-16 years. The aim is to quantitatively explore preliminary effects and qualitatively explore parents' experiences of the program. The aim is also to gain knowledge on whether the support received through the internet-based parenting program and chat support in the program with a family guide (psychologist) is perceived as sufficient, or if additional digital/phone-based meetings with a family guide (psychologist) are more effective and perceived as more helpful.

Research questions are the following:

1. What is the preliminary effect of the internet-based parenting program on children's behavioral problems, emotional and general well-being, parents' emotion regulation, parenting strategies, and family conflicts?
2. What is the level of parents' engagement in the parenting program, i.e., how many modules, exercises, homework tasks are completed, how much time does it take to complete the program, and what is the dropout rate?
3. Do parents perceive that they learn relevant strategies, that the parenting program is effective, acceptable, useful, and how is the collaboration with the family guide perceived? Do parents experience any adverse effects?
4. Is there any difference in the experience and satisfaction with the program, collaboration with the family guide, parents' motivation, dropout rate, completion of exercises, homework tasks, or trends in the effectiveness of the parenting program, depending on whether additional digital/phone-based meetings with the family guide are also included?

METHOD:

This is a small randomized controlled pilot study based on a mixed-methods approach. Evaluation is conducted using repeated measurements and both within- and between-group comparisons.

Parents from various parts of Sweden can participate. The study is advertised, and parents are informed about the study on a website and can contact the responsible researchers for more information. Both caregivers have to give written informed consent to participate. When parents are interested in participating, inclusion and exclusion criteria are reviewed in a telephone call. Included families are randomized to receive either (1) Internet-based parenting program with support from a family guide via chat function, or (2) The same internet-based parenting program along with digital/phone meetings with a family guide.

The interventions are evaluated using validated self-report questionnaires distributed online through a secure web-platform before and after the program, as well as through a telephone interview after the intervention with participants willing to participate in these. One or both caregivers can complete the evaluation before and after the parenting program and participate in the qualitative interview. Interviews are recorded and transcribed.

POWER CALCULATION:

The primary aim of this pilot study is to investigate experiences of the parenting program approaches. The quantitative and qualitative data collected about each approach with ten families in each condition, i.e., 20 families in total in a pre-post analysis of quantitative data, are considered sufficient to provide an in-depth understanding and preliminary insight into effects, acceptability, usability, relevance, and effectiveness of the interventions.

ANALYSES:

The qualitative analyses will be conducted using content analysis or thematic analysis. For the quantitative analyses, changes within and between groups will be evaluated using paired t-tests, repeated measures ANOVA, and/or Generalized Linear Mixed Models (GLMM). If needed, non-parametric alternatives will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child aged 8-16 years
* The parent perceives that the child gets angry easily, displays defiant behaviors, or that there are parent-child conflicts at home.
* The parent is able to access information in Swedish (the program is currently only in Swedish).

Exclusion Criteria:

* Parent of a child under 8 years or over 16 years of age
* The child does not currently have angry, aggressive, or defiant behaviors.
* The child has autism, severe depression, suicidal thoughts, psychosis, or an eating disorders.
* The parent does not speak Swedish.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in behavior problems on the Disruptive Behavior Disorder scale (oppositional defiant disorder subscale). | Pre- and post-intervention (after 7 weeks)
  The oppositional defiant disorder subscale of the Disruptive Behavior Disorder scale is used for assessing children's behavioral problems. The subscale includes 8 items, rated on a 4-point scale (0 to 3). The scale sum ranges från 0 to a total maximum sum of 24. A higher score indicates more severe behavior problems.
Mean change from baseline in parenting on the Parenting Children and Adolescents Scale | Pre- and post-intervention (after 7 weeks)
  Subscales: encouragement of positive behaviors, setting limits, proactive parenting behaviors. The 21 items are here scored on a 5-point scale (1 to 5) and the total scale sum ranges from 21 to a maximum of 105, with a higher score indicating more positive parenting.
Mean change from baseline in parenting on the Parenting Children and Adolescents Scale: Impact scale | Pre- and post-intervention (after 7 weeks)
  Each of the 21 items in the Parenting Children and Adolescents Scale also includes a question whether it is experienced as a problem (yes/no). Total scale sum ranges between 0 and 21, with a higher sum indicating larger problems and impact.

SECONDARY OUTCOMES:
Mean change from baseline in child wellbeing on the KIDSCREEN-10 | Pre- and post-intervention (after 7 weeks)
  This instrument evaluates how parents perceive the health and well-being of their child or adolescent. The 10 items are scored on a 5-point scale (1 to 5), and the total maximum sum ranges between 10 and 50, with a higher score indicating greater child wellbeing and health-related quality of life. Additionally, the scale includes an overall question about how the child is feeling in general.
Mean change from baseline in child wellbeing on the Strengths and Difficulties Questionnaire | Pre- and post-intervention (after 7 weeks)
  The Strengths and Difficulties Questionnaire is used to assess mental health through a total difficulties score as well as through the five subscales (peer relationship problems, prosocial behavior, emotional symptoms, hyperactivity/inattention, conduct problems). The items are scored on a 3-point scale (0 to 2), and the total difficulties score is generated by summing all subscales except the prosocial scale. The summary score ranges from 0 to 40 where higher summary scores indicate more severe problems.
Mean change from baseline in emotion regulation on the Difficulties in Emotion Regulation Scale | Pre- and post-intervention (after 7 weeks)
  Parents' general emotion regulation ability will be measured with the Difficulties in Emotion Regulation Scale. The 16 items are scored on a 5-point scale (1 to 5), and the total summary score ranges between 16 and 80, with a higher score indicating larger difficulties with emotion regulation.
Mean change from baseline in parental emotion regulation on the Parent Emotion Regulation Scale | Pre- and post-intervention (after 7 weeks)
  Parents' emotion regulation ability will be measured with Parent Emotion Regulation Scale. The 20 items are scored on a 5-point scale (1 to 5). A total summary score ranges between 20 and 100 where a higher score will indicate better regulation of emotional ability.
Mean change in family warmth | Pre- and post-intervention (after 7 weeks)
  These variables are measured with 5 questions from the Family Check-Up Caregiver Assessment Scale, scored on a 5-point scale (1 to 5). Total maximum score ranges between 5 and 25, with a higher score indicating a more positive relation.
Mean change in family conflicts | Pre- and post-intervention (after 7 weeks)
  These variables are measured with 3 questions from the Family Check-Up Caregiver Assessment Scale, scored on a 7-point scale (0 to 6). Total maximum score ranges between 0 and 18, with a higher score indicating larger degree of conflicts.
Mean change in parental satisfaction with the week | From baseline to post-intervention (after 7 weeks). Completed once a week when a new program module is accessed.
  Three questions scored 0 to 10 about parents' satisfaction with the week, with how they have been able to support their child and manage conflicts. Total maximum score ranges between 0-30, with a higher score indicating higher satisfaction.
Parental experiences of the internet-based parenting program explored through qualitative interviews | Interviews are conducted after the internet-based parenting program is completed, between 7 to 12 weeks after the initiation of the program
  Qualitative interviews will explore parents' experiences of participating in and applying the internet-based parenting program, and includes questions about experienced effectiveness, feasibility, satisfaction with the program, level of contentment, acceptance, and relevance of the program. The interviews are partly based on an established scale, modified for this purpose, and self-constructed questions.
Parental experiences of each module in the internet-based parenting program | From baseline to post-intervention (after 7 weeks). Completed once a week after working with a new module.
  Four questions after each module about how the parent experiences the online module and exercises. Rated on a scale 0-10, with a maximum total score ranging between 0 and 40. A higher score indicates greater satisfaction with the module.
Parental experiences of the whole internet-based parenting program | Post-intervention (after 7 weeks)
  Six final questions about the program satisfaction, relevance, and usefulness of the intervention and collaboration with the family guide. Rated between 0-10 with a maximum total score ranging between 0-60. A higher score indicates greater satisfaction with the program.
Parental use of the internet-based parenting program: homework tasks, exercises | From pre- to post-intervention (measured after 7 weeks)
  A summary of the mean number of homework tasks, exercises, modules completed in the program.
Parental use of the internet-based parenting program: time spent working with the program | From pre- to post-intervention (measured after 7 weeks)
  A summary of the mean time spent working with the program (hours, total number of weeks).
Parental use of the internet-based parenting program: drop out rate | From baseline to post intervention (measured after 7 weeks)
  The drop out from the program (number of participants).

OTHER OUTCOMES:
Background information | Pre-intervention
  Parents are asked for concise demographic information about themselves (e.g., age, education) and their child (e.g., age, gender, school grade). A total of 8 questions.
Working alone or with partner in the parenting program | Post-intervention (after completion of the final module, 5-7 weeks after baseline)
  Parents are asked if they have worked alone, with a partner, or another family member or friend.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Enebrink, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No